CLINICAL TRIAL: NCT04167462
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Phase 3 Study to Evaluate the Efficacy and Safety of BMS-986165 in Subjects With Moderate-to-Severe Plaque Psoriasis
Brief Title: An Investigational Study to Evaluate Experimental Medication BMS-986165 Compared to Placebo in Participants With Plaque Psoriasis (POETYK-PSO-3) in Mainland China, Taiwan, and South Korea
Acronym: POETYK-PSO-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM011-065
Record Dates: First submitted 2019-11-15; First posted 2019-11-18 (Actual); Results first posted 2022-11-02 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A:BMS-986165 oral administration (Experimental)
  Interventions: Drug: BMS-986165
- Arm B: Placebo oral administration (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986165 — Specified dose on Specified Days
  Arms: Arm A:BMS-986165 oral administration
Other: Placebo — Specified dose on Specified days
  Arms: Arm B: Placebo oral administration

SUMMARY:
The purpose of this study is to investigate the experimental medication BMS-986165 compared to placebo in participants with moderate to severe plaque psoriasis in mainland China, Taiwan, and South Korea

ELIGIBILITY:
Inclusion Criteria:

* Plaque psoriasis for at least 6 months
* Moderate to severe disease
* Candidate for phototherapy or systemic therapy

Exclusion Criteria:

* Other forms of psoriasis
* History of recent infection
* Prior exposure to BMS-986165

Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2022-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (34):
- China (16):
  - Local Institution - 0001, Beijing, Beijing Municipality
  - Local Institution - 0007, Beijing, Beijing Municipality
  - Local Institution - 0014, Beijing, Beijing Municipality
  - Local Institution - 0008, Chongqing, Chongqing Municipality
  - Local Institution - 0011, Wuhan, Hubei
  - Local Institution - 0016, Wuhan, Hubei
  - Local Institution, Changsha, Hunan
  - Local Institution, Nanjing, Jiangsu
  - Local Institution - 0002, Changchun, Jilin
  - Local Institution - 0006, Dalian, Liaoning
  - Local Institution - 0018, Taiyuan, Shan1xi
  - Local Institution - 0012, Jingan, Shanghai Municipality
  - Local Institution, Chengdu, Sichuan
  - Local Institution - 0009, Hangzhou, Zhejiang
  - Local Institution - 0003, Hangzhou, Zhejiang
  - Local Institution - 0004, Hangzhou, Zhejiang
- South Korea (14):
  - Local Institution - 0034, Bucheon-si
  - Local Institution - 0033, Goyang-si
  - Local Institution - 0028, Gwangju
  - Local Institution - 0035, Incheon
  - Local Institution - 0022, Seongnam-si
  - Local Institution - 0037, Seongnam-si
  - Local Institution - 0036, Seoul
  - Local Institution - 0026, Seoul
  - Local Institution, Seoul
  - Local Institution - 0021, Seoul
  - Local Institution - 0020, Seoul
  - Local Institution - 0027, Seoul
  - Local Institution - 0024, Seoul
  - Local Institution - 0023, Suwon
- Taiwan (4):
  - Local Institution - 0029, Kaohsiung City
  - Local Institution - 0031, Taipei
  - Local Institution - 0032, Taipei
  - Local Institution - 0025, Taoyuan District

REFERENCES:
- [Derived] Zhang J, Ding Y, Wang P, Li L, Pan W, Lu Y, Cheng H, Jiang X, Ho JC, Guo S, Seo SJ, Gold LS, Blauvelt A, Zhuo J, Zhong Y, Becker B, Liu L, Banerjee S, Thaci D. Deucravacitinib, an Oral, Selective, Allosteric Tyrosine Kinase 2 Inhibitor, in Asian Patients With Moderate to Severe Psoriasis: Improvements in Patient-Reported Outcomes in a Randomized Trial. J Dermatol. 2025 Sep;52(9):1360-1367. doi: 10.1111/1346-8138.17834. Epub 2025 Jul 17. PMID 40671612
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: BMS-986165: Participants received a 6 mg tablet of BMS-986165 once daily
- Arm 2: Placebo: Participants received a placebo tablet once daily. After Week 16, participants were transferred to a 6 mg tablet of BMS-986165 once daily
Period: Overall Study
Arm/Group | Arm 1: BMS-986165 | Arm 2: Placebo
Started (Started=treated) | 146 | 74
Completed | 132 | 64
Not Completed | 14 | 10
Not completed — Other reasons | 3 | 2
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Adverse Event | 4 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 2: Placebo: Participants received a placebo tablet once daily
- Total: Total of all reporting groups
Arm/Group | Arm 1: BMS-986165 | Arm 2: Placebo | Total
Number analyzed (Participants) | 146 | 74 | 220
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.3 (12.19) | 41.2 (12.33) | 40.6 (12.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 40
  Male | 123 | 57 | 180
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Chinese | 118 | 62 | 180
  Asian - Korean | 28 | 12 | 40

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With sPGA Response of 0 or 1
Description: static Physician Global Assessment (sPGA) 0 or 1 response assessed as a percentage of participants with a sPGA score of 0 or 1 as assessed at week 16 with at least a 2-point improvement from baseline.
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scale, and induration. The sPGA measure determines psoriasis severity at a single point in time (without taking into account the baseline disease condition) as clear (0), almost clear (1), mild (2), moderate (3), or severe (4). A higher score equates to higher severity of disease. The individual scores at each visit will range from 0-4 and will be captured for erythema, induration, and scaling. A total score will also be computed based on the average of the 3 characteristic scores. The average score will be rounded to the nearest whole number and data for this endpoint will be derived from the total average score.
Time Frame: At week 16
Population: All treated participants. Participants missing results at week 16 due to COVID-19 are excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: BMS-986165 | Arm 2: Placebo
Number analyzed (Participants) | 144 | 74
Percentage of participants | 55.6 [47.4 to 63.7] | 6.8 [1.0 to 12.5]
Statistical Analysis 1: Comparison: Arm 1: BMS-986165 vs Arm 2: Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 16.49, 95% CI 2-sided [6.33 to 42.98]

2. Primary Outcome: The Percentage of Participants With PASI 75 Response
Description: Psoriasis Area and Severity Index (PASI) 75 response is an assessment defined as the percentage of participants who experience at least a 75% improvement in PASI score at Week 16 as compared with baseline value. PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions graded on a scale from 0-4 (0= absent symptoms, 1= mild symptoms, 2= moderate symptoms, 3= severe symptoms, 4= very severe symptoms), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. The PASI includes multiple subscores and a final total score. Individual plaque characteristic rating scores are provided for each body region as well as the weighted score. The PASI Total score will be used to assess response to treatment.
Time Frame: At week 16
Population: All treated participants. Participants missing results at week 16 due to COVID-19 are excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: BMS-986165 | Arm 2: Placebo
Number analyzed (Participants) | 144 | 74
Percentage of participants | 68.8 [61.2 to 76.3] | 8.1 [1.9 to 14.3]
Statistical Analysis 1: Comparison: Arm 1: BMS-986165 vs Arm 2: Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 24.29, 95% CI 2-sided [9.60 to 61.46]

3. Secondary Outcome: The Percentage of Participants With PASI 90 Response
Description: Psoriasis Area and Severity Index (PASI) 90 response is an assessment defined as the percentage of participants who experience at least a 90% improvement in PASI score at Week 16 as compared with baseline value. PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions graded on a scale from 0-4 (0= absent symptoms, 1= mild symptoms, 2= moderate symptoms, 3= severe symptoms, 4= very severe symptoms), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. The PASI includes multiple subscores and a final total score. Individual plaque characteristic rating scores are provided for each body region as well as the weighted score. The PASI Total score will be used to assess response to treatment.
Time Frame: At week 16
Population: All treated participants. Participants missing results at week 16 due to COVID-19 are excluded. Pre-specified data collected for Arms 1 and 2 at Week 16.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: BMS-986165 | Arm 2: Placebo
Number analyzed (Participants) | 144 | 74
Percentage of participants | 38.2 [30.3 to 46.1] | 1.4 [0.0 to 4.0]
Statistical Analysis 1: Comparison: Arm 1: BMS-986165 vs Arm 2: Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 41.19, 95% CI 2-sided [5.82 to 291.26]

4. Secondary Outcome: The Percentage of Participants With PASI 100 Response
Description: Psoriasis Area and Severity Index (PASI) 100 response is an assessment defined as the percentage of participants who experience at least a 100% improvement in PASI score at Week 16 as compared with baseline value. PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions graded on a scale from 0-4 (0= absent symptoms, 1= mild symptoms, 2= moderate symptoms, 3= severe symptoms, 4= very severe symptoms), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. The PASI includes multiple subscores and a final total score. Individual plaque characteristic rating scores are provided for each body region as well as the weighted score. The PASI Total score will be used to assess response to treatment.
Time Frame: At week 16
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: BMS-986165 | Arm 2: Placebo
Number analyzed (Participants) | 144 | 74
Percentage of participants | 4.2 [0.9 to 7.4] | 0 [0 to 0]

5. Secondary Outcome: The Percentage of Participants With sPGA 0 Response
Description: static Physician Global Assessment (sPGA) 0 response is defined as the percentage of participants with a sPGA score of 0 with at least 2-point improvement from baseline as assessed at Week 16.
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scale, and induration. The sPGA measure determines psoriasis severity at a single point in time (without taking into account the baseline disease condition) as clear (0), almost clear (1), mild (2), moderate (3), or severe (4). A higher score equates to higher severity of disease. The individual scores at each visit will range from 0-4 and will be captured for erythema, induration, and scaling. A total score will also be computed based on the average of the 3 characteristic scores. The average score will be rounded to the nearest whole number and data for this endpoint will be derived from the total average score.
Time Frame: At week 16
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: BMS-986165 | Arm 2: Placebo
Number analyzed (Participants) | 144 | 74
Percentage of participants | 13.9 [8.2 to 19.5] | 0 [0 to 0]

6. Secondary Outcome: Change From Baseline in PSSD Symptom Score
Description: Change from baseline in Psoriasis Symptoms and Signs Diary (PSSD) symptom score is defined as the percentage of participants with a PSSD score of 0 among participants with a baseline PSSD symptom score ≥ 1.
  The PSSD is an 11-item participant-reported instrument that assesses severity of symptoms and participant-observed signs commonly associated in plaque psoriasis. The PSSD assesses severity of 5 symptoms (itch, pain, stinging, burning, skin tightness) and 6 participant-observed signs (skin dryness, cracking, scaling, shedding or flaking, redness, bleeding) using 0-10 numerical ratings. The severity of each item is rated on an 11-point numeric rating scale ranging from 0 (absent) to 10 (worst imaginable). A symptom score will be derived by averaging the 5 questions and multiplying by 10. A sign score will be derived by averaging the 6 questions and multiplying by 10. A total PSSD score with range 0-100 will be derived from taking the average of the symptom and sign scores.
Time Frame: Baseline and at Week 16
Population: Participants with a baseline PSSD symptom score ≥ 1. Participants missing results at week 16 due to COVID-19 are excluded. Pre-specified data collected for Arms 1 and 2 at Week 16.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm 1: BMS-986165 | Arm 2: Placebo
Number analyzed (Participants) | 142 | 73
Score on a scale | -29.4 (23.21) | -1.8 (25.32)

7. Secondary Outcome: The Percentage of Participants With Ss-PGA Score of 0 or 1
Description: Scalp specific Physician's Global Assessment (ss-PGA) 0 or 1 assessed at Week 16 as a percentage of participants with a ss-PGA score 0 or 1 among participants with a baseline ss-PGA score ≥3.
  The ss-PGA is assessed at each visit throughout the study in participants that have evidence of scalp psoriasis at baseline. If there is evidence of scalp involvement, scalp lesions are evaluated in terms of clinical signs of redness, thickness, and scaliness and scored on the following 5-point ss-PGA scale:
  0 = absence of disease, 1 = very mild disease, 2 = mild disease, 3 = moderate disease, 4 = severe disease.
Time Frame: At week 16
Population: Participants with a baseline ss-PGA score ≥3. Participants missing results at week 16 due to COVID-19 are excluded. Pre-specified data collected for Arms 1 and 2 at Week 16.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: BMS-986165 | Arm 2: Placebo
Number analyzed (Participants) | 105 | 51
Percentage of participants | 62.9 [53.6 to 72.1] | 9.8 [1.6 to 18.0]
Statistical Analysis 1: Comparison: Arm 1: BMS-986165 vs Arm 2: Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 17.27, 95% CI 2-sided [6.06 to 49.25]

8. Secondary Outcome: The Percentage of Participants With DLQI Score of 0 or 1
Description: Dermatology Life Quality Index 0 or 1 assessed at Week 16 as a percentage of participants with a DLQI score of 0 or 1 among participants with a baseline DLQI score ≥2.
  The DLQI is a participant-reported quality of life index which consists of 10 questions concerning symptoms and feelings, daily activities, leisure, work, school, personal relationships, and treatment during the last week. Each question is scored on a scale of 0 to 3 where a higher value signifies higher severity, with 0="not at all", 1="a little", 2="a lot", or 3="very much". The scores are summed, giving a range from 0 (no impairment of life quality) to 30 (maximum impairment). Interpretation of DLQI scores is as follows:
  1. 0-1 = no effect at all on participant's life
  2. 2-5 = small effect on participant's life
  3. 6-10 = moderate effect on participant's life
  4. 11-20 = very large effect on participant's life
  5. 21-30 = extremely large effect on participant's life
Time Frame: At week 16
Population: Participants with a baseline DLQI score ≥2. Pre-specified data collected for Arms 1 and 2 at Week 16.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: BMS-986165 | Arm 2: Placebo
Number analyzed (Participants) | 140 | 69
Percentage of participants | 36.4 [28.5 to 44.4] | 11.6 [4.0 to 19.1]
Statistical Analysis 1: Comparison: Arm 1: BMS-986165 vs Arm 2: Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 5.10, 95% CI 2-sided [2.19 to 11.91]

9. Secondary Outcome: The Percentage of Participants With PGA-F Score of 0 or 1
Description: Physician's Global Assessment of Fingernail Psoriasis (PGA-F) score of 0 or 1 assessed at Week 16 as a percentage of participants with a PGA-F score of 0 or 1 with at least a 2-point improvement from baseline among participants with a baseline PGA-F score ≥3.
  If a participant shows evidence of psoriatic fingernail involvement, the assessment will be performed at each subsequent visit to assess severity and improvement over time. Only participants with a PGA-F score at baseline will be assessed throughout the study. The overall condition of the fingernails is rated on a 5-point scale:
  0 = clear, 1 = minimal, 2 = mild, 3 = moderate, and 4 = severe
Time Frame: At week 16
Population: Participants with a baseline PGA-F score ≥3. Participants missing results at week 16 due to COVID-19 are excluded. Pre-specified data collected for Arms 1 and 2 at Week 16.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: BMS-986165 | Arm 2: Placebo
Number analyzed (Participants) | 46 | 24
Percentage of participants | 19.6 [8.1 to 31.0] | 4.2 [0.0 to 12.2]
Statistical Analysis 1: Comparison: Arm 1: BMS-986165 vs Arm 2: Placebo; Test type: Superiority; p = 0.0947, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 5.86, 95% CI 2-sided [0.64 to 53.28]

10. Secondary Outcome: The Percentage of Participants With PSSD Symptom Score of 0
Description: Psoriasis Symptoms and Signs Diary (PSSD) symptom score of 0 assessed as a percentage of participants with a PSSD symptom score of 0 among participants with a baseline PSSD symptom score ≥1.
  The PSSD is an 11-item participant-reported instrument that assesses severity of symptoms and participant-observed signs commonly associated in plaque psoriasis. The PSSD assesses severity of 5 symptoms (itch, pain, stinging, burning, skin tightness) and 6 participant-observed signs (skin dryness, cracking, scaling, shedding or flaking, redness, bleeding) using 0-10 numerical ratings. The severity of each item is rated on an 11-point numeric rating scale ranging from 0 (absent) to 10 (worst imaginable). A symptom score will be derived by averaging the 5 questions included in the symptom score and multiplying by 10. scores range from 0-100, where 0 representing the least severe symptom and 100 the most severe.
Time Frame: At week 16
Population: Participants with a baseline PSSD symptom score ≥1. Pre-specified data collected for Arms 1 and 2 at Week 16.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: BMS-986165 | Arm 2: Placebo
Number analyzed (Participants) | 142 | 73
Percentage of participants | 4.9 [1.4 to 8.5] | 1.4 [0.0 to 4.0]
Statistical Analysis 1: Comparison: Arm 1: BMS-986165 vs Arm 2: Placebo; Test type: Superiority; p = 0.1741, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.11, 95% CI 2-sided [0.47 to 35.74]

11. Secondary Outcome: The Percentage of Participants With Pp-PGA Score of 0 or 1
Description: Palmoplantar PGA (pp-PGA) 0/1 assessed as a percentage of participants with a pp-PGA score of 0 or 1 among participants with a baseline pp-PGA score ≥3.
  This measure will be used for participants with palmoplantar (finger and toe surfaces) involvement at baseline. Only participants with baseline palmoplantar involvement will continue to have these assessments at each subsequent visit throughout the study. The pp-PGA uses a 5-point (0-4) overall severity scale:
  0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; and 4 = severe.
Time Frame: At week 16
Population: Participants with a baseline pp-PGA score ≥3. Pre-specified data collected for Arms 1 and 2 at Week 16.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: BMS-986165 | Arm 2: Placebo
Number analyzed (Participants) | 15 | 7
Percentage of participants | 66.7 [42.8 to 90.5] | 0 [0 to 0]

12. Secondary Outcome: The Percentage of Participants With PASI 75 Response at Week 52
Description: Psoriasis Area and Severity Index (PASI) 75 response is an assessment defined as the percentage of participants who experience at least a 75% improvement in PASI score at Week 52 as compared with participants that are PASI 75 responders at Week 16. PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions graded on a scale from 0-4 (0= absent symptoms, 1= mild symptoms, 2= moderate symptoms, 3= severe symptoms, 4= very severe symptoms), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. The PASI includes multiple subscores and a final total score. Individual plaque characteristic rating scores are provided for each body region as well as the weighted score. The PASI Total score will be used to assess response to treatment.
Time Frame: At week 52
Population: All treated participants. Data is represented from participants original randomization arm.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: BMS-986165 | Arm 2: Placebo
Number analyzed (Participants) | 145 | 74
Percentage of participants | 71.0 [63.7 to 78.4] | 70.3 [59.9 to 80.7]

13. Secondary Outcome: The Percentage of Participants With sPGA Response of 0 or 1 at Week 52
Description: static Physician Global Assessment (sPGA) 0 or 1 response assessed as a percentage of participants with a sPGA score of 0 or 1 as assessed at week 52 among participants that are sPGA 0 or 1 responders at Week 16.
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scale, and induration. The sPGA measure determines psoriasis severity at a single point in time (without taking into account the baseline disease condition) as clear (0), almost clear (1), mild (2), moderate (3), or severe (4). A higher score equates to higher severity of disease. The individual scores at each visit will range from 0-4 and will be captured for erythema, induration, and scaling. A total score will also be computed based on the average of the 3 characteristic scores. The average score will be rounded to the nearest whole number and data for this endpoint will be derived from the total average score.
Time Frame: At week 52
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: BMS-986165 | Arm 2: Placebo
Number analyzed (Participants) | 145 | 74
Percentage of participants | 51.0 [42.9 to 59.2] | 52.7 [41.3 to 64.1]

ADVERSE EVENTS:
Time Frame: SAEs and NSAEs: From first dose to 100 days post last dose (up to approximately 15 months). All-Cause Mortality: From first dose through the course of the trial (up to approximately 24 months).
Groups:
- Placebo Week 0 up to Week 16: Participants received a placebo tablet once daily from Week 0 up to Week 16
- BMS-986165 Week 0 up to Week 52: Participants received a 6 mg tablet of BMS-986165 once daily from Week 0 up to Week 52
- BMS-986165 Week 16 up to Week 52: Participants from the placebo group were switched to receive a 6 mg tablet of BMS-986165 once daily from Week 16 up to Week 52.
Arm/Group | Placebo Week 0 up to Week 16 | BMS-986165 Week 0 up to Week 52 | BMS-986165 Week 16 up to Week 52
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/146 | 0/68
Serious Adverse Events (participants affected / at risk) | 3/74 | 4/146 | 0/68
Other Adverse Events (participants affected / at risk) | 29/74 | 55/146 | 19/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Week 0 up to Week 16 (N=74) | BMS-986165 Week 0 up to Week 52 (N=146) | BMS-986165 Week 16 up to Week 52 (N=68)
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis shigella (Infections and infestations) | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hepatobiliary procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cyst (General disorders) | 1 | 0 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Week 0 up to Week 16 (N=74) | BMS-986165 Week 0 up to Week 52 (N=146) | BMS-986165 Week 16 up to Week 52 (N=68)
Mouth ulceration (Gastrointestinal disorders) | 4 | 11 | 0
Nasopharyngitis (Infections and infestations) | 6 | 10 | 4
Upper respiratory tract infection (Infections and infestations) | 14 | 26 | 4
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4
Headache (Nervous system disorders) | 0 | 8 | 4
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 4 | 8
Folliculitis (Infections and infestations) | 4 | 5 | 1
Pharyngitis (Infections and infestations) | 4 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT04167462/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT04167462/SAP_001.pdf